CLINICAL TRIAL: NCT00518557
Title: Combination Treatment of TACE With Recombinant Human Endostatin Administrated Via Hepatic Artery in Hepatocellular Carcinoma
Brief Title: Synergistic Treatment for Hepatocellular Carcinoma (HCC) Using TACE With Antiangiogenesis
Acronym: TACE HCC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Southeast University, China (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SIMCERE-123456
Record Dates: First submitted 2007-08-16; First posted 2007-08-20 (Estimated); Last update posted 2009-01-22 (Estimated); Status verified 2009-01

CONDITIONS: Hepatocellular Carcinoma
Keywords: liver cancer; interventional radiology; Chemoembolization; Safety; Effectiveness
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): All patients of this arm are treated by TACE together with Andostatin.
  Interventions: Procedure: Transcatheter Arterial Chemoembolization
- 2 (Active Comparator): All patients of this arm are treated by TACE alone: only mixture of Epirubicin and Lipiodol is injected into the feeding arteries of the tumor, without injection of Andostatin.
  Interventions: Procedure: Transcatheter Arterial Chemoembolization

INTERVENTIONS:
Procedure: Transcatheter Arterial Chemoembolization — The interventional procedure is performed as following steps: 1)transcatheter hepatic arterial angiography(including any feeding arteries to the tumor) is performed under a DSA unit; 2) super selectively catheterizaton of feeding arteries to the tumor is reached; 3)30 mg of Andostatin (Simcere Co. China) mixtured with 5 ml Lipiodol is injected into the tumor via the feeding arteries; 4) followed by 10 mg of Epifubicin mixtured with 5 ml of Lipiodol; 5) All feeding arteries to the tumor are occluded which is confirmed by re-angiography.
  Other Names: TAE

SUMMARY:
The purpose of this study is to investigate safety and potential therapeutic benefits for patients with hepatocellular carcinoma by transcatheter chemoembolization with the recombinant endostatin (commercially available in China)which is also administrated via the hepatic artery. The hypothesis of this protocol is that TACE with antiangiogenic treatment may inhibit the proangiogenic effects induced by the hypoxia of TACE.

ELIGIBILITY:
Inclusion Criteria:

* Patients with cytologically or histologically documented HCC, who are candidates for TACE
* Child-Pugh Child A or B
* Age >= 18
* Measurable disease by RECIST criteria;
* Performance status ECOG 0-2
* Previous local therapy completed > 4 weeks
* Written informed consent signed
* Normal organ and marrow function defined as:

Haematopoietic:

* WBC ≥ 3,000/µlplatelet count > 80,000/mm3
* haemoglobin > 9g/dL
* Hepatic: Albumin ≥ 2.8 g/dl.serum total bilirubin ≤ 3 mg/dl; AST or ALT < 5 x ULN
* Renal: creatinine < 1.5 x ULN

Exclusion Criteria:

* Metastases
* Prior or concomitant chemotherapy or radiation therapy
* VEGF/VEGFR- inhibitors or other anti-angiogenesis agents
* Severe and/or uncontrolled medical conditions:
* Congestive heart failure, serious cardiac arrhythmia, active coronary artery
* Severe renal impairment
* Patients who anticipate receiving major surgery during the course of the
* Pregnant or breastfeeding patients
* Evidence of bleeding diathesis

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2007-04; Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability, Mortality | 6 months

SECONDARY OUTCOMES:
Tumor volumetry, Changes of Tumor markers such as AFP, Curriculum survival | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Gao-Jun Teng, MD, Ph.D, Principal Investigator — Zhongda Hospital, Southeast University, Nanjing, China
Locations (1):
- Department of Interventional Radiology, Zhongda Hospital, Southeast University, Nanjing, Jiangsu, China

REFERENCES:
- See also: Related Info — http://www.ncbi.nlm.nih.gov